CLINICAL TRIAL: NCT06901453
Title: Effectiveness of RMGI and Giomer, Both Individually and in Combination, for Restoring Anterior Cervical Caries in High-Risk Patients: A Randomized Clinical Trial
Brief Title: The Effectiveness RMGI and Giomer, Individually and Combined Anterior Cervical Caries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Magdy Eldamanhoury, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoU-Bioactive Veneering
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Cervical Caries
Keywords: Risk Factor; Patient Outcome Assessment
MeSH Terms: conditions — Dental Caries; Root Caries

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial compares three bioactive restorative materials (Giomer, RMGI veneered with Giomer, and RMGI alone) for treating anterior cervical caries in high-risk patients. 75 participants (25 per group) will be evaluated over 18 months for secondary caries (primary outcome), restoration integrity, appearance, and sensitivity using modified USPHS criteria at baseline, 6, 12, and 18 months. The parallel-group superiority design with 1:1:1 allocation will include blinded outcome assessment at the Conservative Dentistry Department, Cairo University.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors (A.Y. & D.E.), who are experienced clinicians responsible for evaluating the restorations at each follow-up period (baseline, 6, 12, and 18 months), are kept completely unaware of which treatment each patient received. They evaluate all restorations using standardized criteria without knowledge of the group allocation. Additionally, the statistician who analyzes the collected data is also blinded to the treatment groups during the statistical analysis process, ensuring unbiased interpretation of results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 2 (RMGI + Giomer Lamination) (Experimental): Cavities will be restored using a combination technique where light-cured resin modified glass ionomer (GC Fuji II LC) is applied first, leaving 1.5mm space for Giomer. After selective enamel etching, adhesive will be applied to both enamel and dentin margins as well as the RMGI floor, followed by application of Beautifil II LS Giomer as the final layer.
  Interventions: Procedure: RMGI alone - Control
- Group 3 (RMGI alone - Control) (Active Comparator): Cavities will be restored with light-cured resin modified glass ionomer (GC Fuji II LC) only. After applying conditioner for 20 seconds, rinsing, and gentle drying, the RMGI will fill the entire cavity and be light-cured. GC Fuji Varnish will be applied before and after finishing to prevent moisture penetration.
  Interventions: Procedure: Low shrinkage Giomer restorative material (Beautifil II LS)
- Group 1 (Giomer) (Active Comparator): Cavities will be restored with low shrinkage Giomer restorative material (Beautifil II LS, Shofu, Japan). After etching enamel margins with 37% phosphoric acid for 15 seconds, FL bond two-step self-etch adhesive will be applied, followed by incremental application of Giomer (maximum 2mm thickness) with light-curing for 20 seconds.
  Interventions: Procedure: RMGI alone - Control

INTERVENTIONS:
Procedure: Low shrinkage Giomer restorative material (Beautifil II LS) — Enamel margins are etched with 37% phosphoric acid for 15 seconds, then the cavity is bonded using FL bond two-step self-etch adhesive. Giomer is applied in increments (maximum 2mm thickness) and light-cured for 20 seconds with a properly calibrated LED curing light.
  Arms: Group 3 (RMGI alone - Control)
Procedure: RMGI alone - Control — Cavities will be restored with light-cured resin modified glass ionomer (GC Fuji II LC) only. After applying conditioner for 20 seconds, rinsing, and gentle drying, the RMGI will fill the entire cavity and be light-cured
  Arms: Group 1 (Giomer); Group 2 (RMGI + Giomer Lamination)

SUMMARY:
This study compares the effectiveness of three dental materials for restoring anterior cervical caries in high-risk patients: resin-modified glass ionomer (RMGI), Giomer, and a combination technique where RMGI is veneered with Giomer. The 18-month randomized clinical trial will assess 75 patients (25 per group), primarily evaluating secondary caries formation, with additional measurements of restoration integrity, appearance, and sensitivity at baseline, 6, 12, and 18 months.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical performance of three different restorative materials for treating anterior cervical caries in high-risk patients over 18 months. The research will compare resin-modified glass ionomer (RMGI), Giomer, and a combination technique where RMGI is veneered with Giomer (lamination technique). The randomized controlled clinical trial will involve 75 patients, with 25 patients in each treatment group. The primary outcome is secondary caries assessment, while secondary outcomes include fracture, retention, marginal integrity, marginal discoloration, anatomic form, surface texture, and postoperative sensitivity. Assessments will occur at baseline, 6, 12, and 18 months using modified USPHS criteria.

The rationale behind this study is that high-risk caries patients need restorative materials that provide both protection against recurrent decay and aesthetic outcomes. The bioactive properties of these materials, including fluoride release and remineralization capabilities, make them potentially suitable for these patients. The research protocol includes detailed methods for patient selection, randomization, blinding, treatment procedures, follow-up assessments, and statistical analysis. The study is self-funded and will be conducted at the Conservative Dentistry Department, Faculty of Dentistry, Cairo University, with appropriate ethical approvals and informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patient age range from 18-55 years
* Presence of anterior cervical caries on the labial surface (ICDAS 4 & 5)
* High caries risk
* Good general health

Exclusion Criteria:

* Severe or chronic periodontal disease
* Bruxism
* Non-vital teeth
* Fractured or cracked teeth
* Defective restorations
* Pregnancy and/or lactation
* Allergy to the main components of the products to be used in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Secondary Caries | 6 months
  The methodology includes visual examination, short air drying, and the use of a 250-μm probe to assess for the presence of secondary caries around the restorations.
Secondary Caries | 12 months
  The methodology includes visual examination, short air drying, and the use of a 250-μm probe to assess for the presence of secondary caries around the restorations.
Secondary Caries | 18 months
  The methodology includes visual examination, short air drying, and the use of a 250-μm probe to assess for the presence of secondary caries around the restorations.

IPD SHARING:
Plan to Share IPD: No